CLINICAL TRIAL: NCT00932828
Title: Determining the Efficacy and Value of Immunotherapy on the Likelihood of Peanut Tolerance: The DEVIL Study; Grant "Optimizing Tolerance Induction in Peanut Allergy: The DEVIL Study"
Brief Title: Determining the Efficacy and Value of Immunotherapy on the Likelihood of Peanut Tolerance: The DEVIL Study
Acronym: DEVIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2307
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-02

CONDITIONS: Food Hypersensitivity
Keywords: Peanut allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: For the purposes of the primary outcome, all subjects will receive peanut OIT and represent a single group. For exploratory analysis, subjects will be randomized to high and low dose OIT to potentially look for a dose response.
Masking Description: For exploratory analysis, subjects will be randomized 1:1 to high (3000mg) and low dose (300mg) OIT to potentially look for a dose response. Low dose will be masked by adding oat flour to provide a dose equal to high dose with respect to flour but with lower peanut protein content
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peanut oral immunotherapy (Experimental): Newly diagnosed allergic children receiving peanut flour as oral immunotherapy for the treatment of peanut allergy.
  Interventions: Drug: Peanut oral immunotherapy

INTERVENTIONS:
Drug: Peanut oral immunotherapy — Defatted peanut in flour form to be used as treatment for peanut allergy
  Other Names: Peanut mucosal immunotherapy; Peanut OIT

SUMMARY:
Peanut allergy is known to cause severe anaphylactic reactions.The goal of this proposal is to produce a new treatment that would benefit young subjects who have recently been diagnosed with peanut allergy by lowering the risk of anaphylactic reactions (desensitization), and changing the peanut-specific immune response in subjects who have peanut allergy (tolerance).

DETAILED DESCRIPTION:
Peanut allergy is known to cause severe anaphylactic reactions. Compared with other food allergies, it tends to be more persistent and its prevalence seems to be rising. Currently, there is no proven treatment other than strict avoidance. We are attempting to decrease the risk of anaphylaxis on accidental ingestion by desensitizing subjects to peanut using peanut mucosal immunotherapy (PMIT) more commonly called oral immunotherapy (OIT). We are also studying the effect of PMIT on the peanut-specific immune response to determine if tolerance to peanut protein will develop. Based on our preliminary work and recent studies supporting the importance of early oral exposure in tolerance induction, we propose that early treatment of peanut allergy with PMIT will be safe and effective. Children ages 9 to 36 months with peanut allergy will be randomized to receive high or low dose PMIT using peanut flour. Subjects will undergo desensitization on the first day and then increase the doses gradually to a maintenance dose. Doses will be taken daily at home except for dose increases which will be done on the research unit. Subjects will undergo a double-blinded, placebo-controlled food challenge (DBPCFC) if challenge criteria are met. Subjects passing the first challenge will stop PMIT and repeat the DBPCFC to assess tolerance. Outcome variables of interest include response to oral food challenges (OFC), skin prick testing, peanut specific serum immunoglobin E (IgE), immunoglobin G (IgG), and immunoglobin G4 (IgG4) and stool immunoglobin A (IgA), T and B cell responses, quality of life, and adverse events. As secondary and exploratory outcomes, these longitudinal results will be compared between high and low dose PMIT groups and controls using appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 9-36 months of either sex, any race, any ethnicity at the time of the initial visit
* EITHER a positive skin prick test to peanuts or in vitro [CAP-FEIA] peanut immunoglobin E (IgE) level in the blood > 0.35 kU/L PLUS a history of a clinical allergic reaction (defined as significant clinical symptoms occurring within 60 minutes after ingesting peanuts) within 6 months of screening
* OR a positive prick skin test to peanuts and in vitro [CAP-FEIA] peanut IgE level > 5 kU/L when there is no history of allergic reaction and no known peanut exposure
* Provision of signed informed consent
* Development of symptoms characteristic of IgE-mediated food allergy (urticaria, angioedema, respiratory distress/wheeze/cough, vomiting/diarrhea, anaphylaxis) during initial oral food challenge

Exclusion Criteria:

* History of severe anaphylaxis to peanut as defined by hypoxia, hypotension, or neurological compromise
* Currently participating in a study using an investigational new drug
* Participation in any interventional study for the treatment of food allergy in the past 12 months
* Subjects with a known wheat food allergy will be excluded because of cross contamination of oat with wheat
* Severe atopic dermatitis
* Currently being treated with greater than medium daily doses of inhaled corticosteroids, as defined by the National Heart Lung and Blood Institute (NHLBI) guidelines
* Inability to discontinue antihistamines for skin testing and OFCs

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-06-22 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvil W Burks, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vickery BP, Berglund JP, Burk CM, Fine JP, Kim EH, Kim JI, Keet CA, Kulis M, Orgel KG, Guo R, Steele PH, Virkud YV, Ye P, Wright BL, Wood RA, Burks AW. Early oral immunotherapy in peanut-allergic preschool children is safe and highly effective. J Allergy Clin Immunol. 2017 Jan;139(1):173-181.e8. doi: 10.1016/j.jaci.2016.05.027. Epub 2016 Aug 10. PMID 27522159

RESULTS

PARTICIPANT FLOW:
Groups:
- Peanut Oral Immunotherapy: All subjects are treated with peanut oral immunotherapy for primary outcome. Patients randomized to 300mg or 3000mg for secondary dose finding outcome.
Period: Overall Study
Arm/Group | Peanut Oral Immunotherapy
Started | 37
Completed | 32 (5 subjects who did not complete the protocol were considered in an ITT analysis.)
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Peanut Oral Immunotherapy: All subjects who are treated with peanut OIT (300mg or 3000mg) and undergo a DBPCFC after 36 months of treatment and an additional DBPCFC after 4 weeks of treatment avoidance. Analysis was completed ITT.
Arm/Group | Peanut Oral Immunotherapy
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 28.5 [22 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37
Peanut immunoglobin E (IgE) [Median (Inter-Quartile Range); unit: kUA/L] | 14.4 [3.4 to 48.6]
Peanut skin prick test (SPT) [Median (Inter-Quartile Range); unit: mm wheal size] — Epicutaneous skin prick test applied using the Greer pick and measured after 15 minutes. Cross diameters of the raised wheal skin response are averaged and reported as the average wheal size in mm.
  mm wheal size | 11.5 [8 to 16.5]

OUTCOME MEASURES:

1. Primary Outcome: Determine the Percentage of Subjects Who Demonstrate Sustained Unresponsiveness (SU) by a Negative Double-blind Placebo-controlled Food Challenge (DBPCFC).
Description: The goal of the study is to treat peanut-allergic subjects with peanut OIT and to determine whether this protocol lowers their risk of anaphylactic reactions and causes SU. We expect to demonstrate the effectiveness of peanut OIT in inducing SU by showing that subjects will have a negative DBPCFC to 5 grams of peanut following completion of a 36-month course of peanut OIT followed by avoidance of therapy for 4 weeks.
Time Frame: After 36 months of OIT dosing followed by 1 month of avoidance
Population: 37 subjects considered with ITT analysis including 5 withdrawals
Measure: Count of Participants; unit: Participants
Groups:
- Peanut Oral Immunotherapy: All subjects who are treated with peanut OIT (300mg or 3000mg) and undergo a DBPCFC after 36 months of treatment and an additional DBPCFC after 4 weeks of treatment avoidance. Analysis was completed as ITT.
Arm/Group | Peanut Oral Immunotherapy
Number analyzed (Participants) | 37
Participants | 29

2. Secondary Outcome: Determine the Percentage of Subjects Who Demonstrate Desensitization by a Negative Double-blind Placebo-controlled Food Challenge (DBPCFC).
Description: We expect to demonstrate the effectiveness of peanut OIT in inducing desensitization by showing that subjects will have a negative DBPCFC to 5 grams of peanut following completion of a 36-month course of peanut OIT .
Time Frame: After 36 months of OIT dosing
Population: 37 subjects considered with ITT analysis including 5 withdrawals
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Oral Immunotherapy
Number analyzed (Participants) | 37
Participants | 30

3. Secondary Outcome: Determine the Frequency of Treatment-related Adverse Effects (TAE) From Peanut OIT.
Description: In addition to studying the effectiveness of peanut OIT, we will also determine the safety of peanut OIT by reporting the average rate of TAEs per person per dose.
Time Frame: After 36 months of OIT dosing followed by 1 month of avoidance
Population: 37 subjects considered with ITT analysis including 5 withdrawals
Measure: Median (95% Confidence Interval); unit: AEs per person per dose
Arm/Group | Peanut Oral Immunotherapy
Number analyzed (Participants) | 37
AEs per person per dose | 0.8 [0.3 to 1.4]

ADVERSE EVENTS:
Time Frame: TAEs reported over the course of 36 months of peanut OIT treatment for each subject
Arm/Group | Peanut Oral Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 35/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peanut Oral Immunotherapy (N=37)
Abdominal pain (Gastrointestinal disorders) | 22
Skin/oral pruritus (Skin and subcutaneous tissue disorders) | 19
Nausea/vomiting (Gastrointestinal disorders) | 23
Sneezing/congestion (Respiratory, thoracic and mediastinal disorders) | 13
Hives (Skin and subcutaneous tissue disorders) | 20
Rash (not hives) (Skin and subcutaneous tissue disorders) | 29
Multiple symptoms (General disorders) | 11 — Multiple symptoms included any single reaction that involved multiple systems (skin/gastrointestinal/upper respiratory/lower respiratory). This group does not overlap with the other groups that involved isolated symptoms in each specified category.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-04-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT00932828/Prot_000.pdf
  • Statistical Analysis Plan (2013-04-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT00932828/SAP_001.pdf